CLINICAL TRIAL: NCT02741843
Title: Impact of Patient Education on Influenza Vaccine Uptake Among Community-dwelling Chinese Elderly: A Randomised Controlled Trial
Brief Title: Impact of Patient Education on Influenza Vaccine Uptake Among Community-dwelling Chinese Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Purpose: Health Services Research
Other Study IDs: HKUCTR-1930
Record Dates: First submitted 2016-04-13; First posted 2016-04-18 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-05

CONDITIONS: Influenza, Human
MeSH Terms: conditions — Influenza, Human | interventions — Patient Education as Topic

ARMS (2):
- Patient Education (Experimental)
  Interventions: Behavioral: Patient Education
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Patient Education
  Arms: Patient Education

SUMMARY:
The purpose of this study is to test the effectiveness of brief face-to-face patient education in increasing uptake of influenza vaccine among Chinese elderly in the community.

ELIGIBILITY:
Inclusion Criteria:

* Cantonese speaking
* Chinese

Exclusion Criteria:

* cognitively impaired
* unable to communicate effectively
* having known contraindication of vaccination
* institutionalized

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Dates: Start 2015-10; Primary Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
proportion of patients receiving influenza vaccination | three working days

SECONDARY OUTCOMES:
proportion of patients receiving influenza vaccination | five working days
proportion of patients receiving influenza vaccination | seven working days
proportion of patients receiving influenza vaccination | nine working days

REFERENCES:
- [Derived] Leung KC, Mui C, Chiu WY, Ng YY, Chen MHY, Ho PH, Kwok CP, Lam SSM, Wong CY, Wong KY, Pang HH. Impact of patient education on influenza vaccine uptake among community-dwelling elderly: a randomized controlled trial. Health Educ Res. 2017 Oct 1;32(5):455-464. doi: 10.1093/her/cyx053. PMID 28931164